CLINICAL TRIAL: NCT03694860
Title: Rapid Sequence Induction in EU: Electronic Survey
Brief Title: Rapid Sequence Induction EU: Electronic Survey (RSIEU)
Acronym: RSIEU
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: European Society of Anaesthesiology (ESA) (Unknown)
Responsible Party: Principal Investigator, Petr Štourač, MD, Doc.MD.Ph.D, Brno University Hospital
Other Study IDs: RSI 2018 EU
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Rapid Sequence Induction
Keywords: crush induction, RSI
MeSH Terms: conditions — Cumulative Trauma Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — Members of European society of anaesthesiology care will obtain an electronic survey considering their clinical practice in RSI
  Other Names: electronic survey

SUMMARY:
Rapid sequence induction (RSI) is a common part of routine anesthesiology practice. However several steps of RSI are not based on evidence based data (EBM) and are considered controversial. In an electronic evaluation form that will be send to European Society of Anaesthesiology (ESA) members. The electronic survey will contain 22 question (11 for adult RSI and 11 for paediatric RSI). In the questionnaire the participants will have to describe their routine clinical practice in performing rapid sequence induction.

DETAILED DESCRIPTION:
Rapid sequence induction (RSI) is a common part of routine anesthesiology practice. However several steps of RSI are not based on evidence based data (EBM) and are considered controversial. In an electronic evaluation form that will be send to European Society of Anaesthesiology (ESA) members. The electronic survey will contain 22 question (11 for adult RSI and 11 for paediatric RSI). In the questionnaire the participants will have to describe their routine clinical practice in performing rapid sequence induction.

The 11 will be consulted with the research committee of ESA.

ELIGIBILITY:
Inclusion Criteria:

- Members of European Society of Anaesthesiology

Exclusion Criteria:

- not members of ESA

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Members of Europen Society of Anaesthesiology
Sampling Method: Non-Probability Sample
Enrollment: 1921 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
RSI practice in European countries - questionnaire (electronic survey) | 2 months
  Evaluation of the clinical practice of the RSI European countries

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, doc.MD.Ph.D, Study Chair — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Klucka J, Kosinova M, Zacharowski K, De Hert S, Kratochvil M, Toukalkova M, Stoudek R, Zelinkova H, Stourac P. Rapid sequence induction: An international survey. Eur J Anaesthesiol. 2020 Jun;37(6):435-442. doi: 10.1097/EJA.0000000000001194. PMID 32221099